CLINICAL TRIAL: NCT05763498
Title: Uterine Junctional Zone Evaluation on 3D Ultrasound and Its Relation to Major Adverse Obstetrical Outcomes in Assisted Reproductive Technology
Brief Title: Uterine Junctional Zone and Its Relation to Adverse Obstetrical Outcomes in Assisted Reproductive Technology
Status: Recruiting | Type: Observational
Sponsor: Centro Hospitalar Lisboa Norte (Other)
Responsible Party: Principal Investigator, Isabel Pereira, M.D., Centro Hospitalar Lisboa Norte
Other Study IDs: JZ OO
Record Dates: First submitted 2023-02-27; First posted 2023-03-10 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Infertility, Female
Keywords: infertility; 3D ultrasound; junctional zone
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The junctional zone (JZ) is an internal layer of the myometrium, with unique characteristics that allow its visualization as a hypoechogenic structure in three-dimensional (3D) ultrasound.

While there is a growing realization that the origins of major obstetrical complications associated with defective deep placentation, such as pre-term labour, fetal growth restriction and pre-eclampsia, may lie in the very early pregnancy events, the underlying mechanisms are not understood.

DETAILED DESCRIPTION:
During pregnancy, unique vascular changes occur, associated with decidualization of the maternal tissues in response to trophoblast invasion, first in the endometrium and subsequently in the myometrial JZ. The JZ broadly represents the inner third of the myometrium that, together with its overlying endometrium, is involved in placentation.

Defective deep placentation, defined by the absent or incomplete remodelling of the JZ segment of the spiral arteries, may be associated with a spectrum of obstetrical complications, ranging from late miscarriage and pre-term labour to fetal growth restriction and pre-eclampsia.

Thus, the primary site of vascular pathology in pregnancies lies not in the placenta or decidua but in the JZ. To understand how impaired remodelling of the myometrial JZ prior to conception may predispose to subsequent defective deep placentation, it is important to first describe the structural and functional changes in the JZ at the time of embryo implantation, and subsequently analyse the distinguishing features of defective deep placentation associated with different pregnancy disorders.

Thus, non-invasive assessment of the JZ prior to conception may turn out to be useful in identifying those women at risk of major obstetrical complications.

This project aims to evaluate the relationship between the characteristics of the ZJ in 3D ultrasound, and major adverse obstetrical outcomes in assisted reproductive technology (ART) treatments, namely in vitro fertilization cycles, intracytoplasmic sperm injection and frozen embryo transfer (FET).

In a prospective and observational study with the inclusion of 200 cases, a 3D ultrasound will be performed on the day on which the final oocyte maturation is triggered or, on FET, on the day prior to the administration of progesterone.

After the quality of visualization of the JZ is classified, its thickness will be measured and described as regular, irregular or interrupted.

The volume of the ZJ will be obtained by subtracting the endometrial volume from the volume of the junctional zone and the endometrium.

These characteristics will be related to major obstetrical adverse outcomes: pre-eclampsia, pre-term labour and fetal growth restriction. The relation with a high-risk first trimester screening for pre-eclampsia will also be accessed.

After explaining the study and obtaining written consent, a 3D ultrasound will be performed for uterine evaluation, on the day of the final oocyte maturation trigger in cases of IVF / ICSI. In cases of FET, the ultrasound evaluation will be carried out on the day before the start of the luteal phase support.

All ultrasounds will be performed in a standardized manner by the same operator. With an empty bladder, in a lithotomy position, a 2D transvaginal ultrasound will be performed using a GE Voluson 730 Expert® ultrasound, with an endovaginal probe with a 4-8MHz frequency. Identification of endometriosis lesions or acquired uterine abnormalities such as leiomyomas or adenomyosis will be exclusion criteria. After evaluating the number and maximum dimension of the ovarian follicles and the endometrial thickness, the three-dimensional volume box will be placed to encompass the entire uterus in longitudinal section, with minimal inclusion of para-uterine structures. A maximum acquisition angle of 90º and maximum quality will be used. To minimize artifacts, during the acquisition both the probe and the woman must remain immobile, being asked to hold their breath. Then, a three-dimensional volume will be generated by automatic 360º rotation of the transducer. For each case, two volumes will always be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Women followed in the infertility clinic aged between 18 and 42 years in cycles of IVF, ICSI or endometrial preparation for frozen embryo transfer

Exclusion Criteria:

* Myomas
* adenomyosis
* endometriosis

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Women included are followed in the fertility clinic aged between 18 and 40 years in cycles of IVF, ICSI or endometrial preparation for frozen embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Pre-eclampsia | 40 weeks
  Pre-eclampsia rate
pre-term labour | 37 weeks
  pre-term labour rate
Fetal growth restriction | 40 weeks
  Fetal growth restriction rate

SECONDARY OUTCOMES:
High-risk first trimester screening for pre-eclampsia | 12 weeks
  High-risk first trimester screening for pre-eclampsia rate

CONTACTS AND LOCATIONS:
Overall Officials: Isabel B Pereira, M.D, Principal Investigator — Centro Hospitalar Lisboa Norte
Locations (3):
- Portugal (3):
  - Hospital Central do Funchal, Funchal, Madeira
  - Departamento de Obstetricia, Ginecologia e Medicina da Reprodução, Lisbon
  - Centro Hospitalar Universitário Lisboa Norte, Lisbon